CLINICAL TRIAL: NCT00676143
Title: A Phase Iii, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Efficacy And Safety Trial Of Bapineuzumab (Aab 001, Eln115727) In Subjects With Mild To Moderate Alzheimer Disease Who Are Apolipoprotein E 4 Carriers
Brief Title: Study Evaluating the Safety and Efficacy of Bapineuzumab in Alzheimer Disease Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated on August 6, 2012, because 2 large Phase 3 studies showed no clinical benefit. This decision was not based on any new safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3133K1-3001; B2521002 (Other: Alias Study Number); 2007-005995-14 (EudraCT Number); NCT00909675 (obsolete NCT alias)
Record Dates: First submitted 2008-05-02; First posted 2008-05-12 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer Disease
Keywords: antibody; immunotherapy
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bapineuzumab 0.5 mg/kg (Experimental)
  Interventions: Drug: bapineuzumab
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bapineuzumab — Bapineuzumab 0.5 mg/kg administered by IV infusion approximately every 13 weeks through week 65.
  Other Names: AAB-001
  Arms: Bapineuzumab 0.5 mg/kg
Drug: placebo — Placebo will be administered by IV infusion approximately every 13 weeks through week 65.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of multiple doses of bapineuzumab in patients with mild to moderate Alzheimer Disease. Patients will receive either bapineuzumab or placebo. Each patient's participation will last approximately 1.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD, with MMSE score of 16-26, and brain MRI consistent with the diagnosis of AD
* Concurrent use of cholinesterase inhibitor or memantine allowed, if stable.
* Caregiver will participate and be able to attend clinic visits with patient.

Exclusion Criteria:

* Significant neurological disease other than AD, or a major psychiatric disorder
* Contraindication to undergo brain MRI (e.g., pacemaker, CSF shunt, or foreign metal objects in the body)
* Woman of childbearing potential

Ages: 50 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2008-01; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (284):
- United States (107):
  - Center for Psychiatric Medicine, Birmingham, Alabama
  - Participant and Clinical Interactions Resources, Birmingham, Alabama
  - UAB Clinical Research Pharmacy-Russell Clinic, Birmingham, Alabama
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Jeffrey S. Gitt, DO, PC, Phoenix, Arizona
  - The Compounding Center, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - AC Institute, Incorporated, Carson, California
  - Collaborative Neuroscience Network, Inc, Long Beach, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Alpine Clinical Research Center, Inc., Boulder, Colorado
  - Associated Neurologists, PC, Boulder, Colorado
  - Mile HIgh Research Center, Denver, Colorado
  - Associated Neurologists of Southern Connecticut, P.C., Fairfield, Connecticut
  - Bendheim Cancer Center, Greenwich, Connecticut
  - Center for Healthy Aging, Greenwich, Connecticut
  - Alzheimer's Disease Research Unit, New Haven, Connecticut
  - Hospital Research Unit, New Haven, Connecticut
  - Investigational Drug Service, New Haven, Connecticut
  - Moshe Hasbani, MD, New Haven, Connecticut
  - Norman S. Werdiger, MD, New Haven, Connecticut
  - MR Research Center, New Haven, Connecticut
  - Yale PET Center, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - JEM Research Institute, LLC, Atlantis, Florida
  - JEM Research Institute, Atlantis, Florida
  - Medical Specialist of the Palm Beaches, Atlantis, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research, LLC, Orlando, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Neurostudies Inc, Port Charlotte, Florida
  - Roskamp Institute, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Dekalb Neurology Associates, LLC/NeuroStudies.net, LLC, Decatur, Georgia
  - Neurostudies.net, Decatur, Georgia
  - NeuroStudies.net, Lawrenceville, Georgia
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Southern Illinois University School of Medicine Department, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Univeristy ADCRP, Boston, Massachusetts
  - General Clincial Research Center (Infusion Location), Boston, Massachusetts
  - IDS Pharmacy (Drug Receipt). Attn:Hyesson Hong, Boston, Massachusetts
  - Neuroscience Research of the Berkshires, Pittsfield, Massachusetts
  - Shields MRI, Russells Mills, Massachusetts
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - University of Michigan Hospital and Health System, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - The Center for Pharmaceutical Research P.C., Kansas City, Missouri
  - Memory Enhancement Center of America, Inc., Eatontown, New Jersey
  - Pharmcare USA, Edison, New Jersey
  - Alzheimer's Research Corp./Merician Institute for Aging, Paterson, New Jersey
  - Neurological Care of Central New York, Liverpool, New York
  - Carolina Neuropsychological Services, Inc, Raleigh, North Carolina
  - Healthsouth Blue Ridge Surgery Center, Raleigh, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Radiology Associates, Raleigh, North Carolina
  - Ohio State University Imaging@Martha Moorehouse, Columbs, Ohio
  - The Ohio State University, Columbs, Ohio
  - The Ohio State University, Columbus, Ohio
  - Summit Research Network(Oregon) Inc., Portland, Oregon
  - Providence Brain Institute, Portland, Oregon
  - Providence Cognitive Assessment Clinic, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Dr. Michael Gabe (Clinic), Silverton, Oregon
  - Abington Memorial Hosptial, Abington, Pennsylvania
  - Abington Neurological Associates, Abington, Pennsylvania
  - Abington Neurological Assoc, Abington, Pennsylvania
  - Andorra MRI of Flourtown, Flourtown, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Investigational New Drug Services, Philadelphia, Pennsylvania
  - University of Pennsylvania-Penn Memory Center, Philadelphia, Pennsylvania
  - UPENN Clinical and Transitional Research Center, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Simpson's Pharmacy, Pawtucket, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Medical University of South Carolina Hospitals and Clinics, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC, Charleston, South Carolina
  - Medical University of South Carolina, North Charleston, South Carolina
  - Texas Neurology, P.A., Dallas, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Integra Clinical Research, San Antonio, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Vista Infusions, San Antonio, Texas
  - Inventive Infusion Solutions, San Antonio, Texas
  - Inventive Infusions Solutions, San Antonio, Texas
  - The Memory Clinic, Bennington, Vermont
  - The Pharmacy, Bennington, Vermont
  - Waisman Center (PET only), Madison, Wisconsin
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
  - Wm S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
  - University of Wisconsin Hospitals and Clinics, Madison, Wisconsin
- Argentina (5):
  - Instituto Medico Congreso, Buenos Aires, Buenos Aires
  - Instituto Medico Congreso, Buenos Aires
  - Cemic University Hospital, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Instituto Kremer, Córdoba
- Australia (9):
  - Gosford Hospital; Pharmacy Dept, Gosford, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Hornsby Kuringai Hospital, Hornsby, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - CDAMS Ballarat Base Hospital, Ballarat, Victoria
  - Heidelberg Repatriation Hospital, West Heidelberg, Victoria
  - Hollywood Hospital; Pharmacy Dept, Nedlands, Western Australia
  - McCusker Alzheimer's Research Foundation, Inc., Nedlands, Western Australia
- Austria (5):
  - Medizinische Universitaet Graz, Graz
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - Allg. Krankenhaus der Stadt Wien, Vienna
  - SZ Sued - Kaiser-Franz-Josef-Spital, Vienna
  - Donauspital, Vienna
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - Az. St. Jan Ruddershove 35, Bruges
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - H.-Hartziekenhuis Roeselare-Menen, Roeselare
- Chile (2):
  - Psicomedica Research Group, Santiago, Chile
  - Especialidades Medicas LyS, Santiago
- University Hospital Center Zagreb, Zagreb, Croatia
- Finland (2):
  - Ita-Suomen Yliopisto, Kuopio
  - University of Turku / CRST, Turku
- France (20):
  - CHU de Dijon, Dijon, France
  - CHU Pellegrin, Bordeaux
  - Hopital neurologique du Pr A. Vighetto, Bron
  - Centre d'Imagerie medicale de Basse Normandie, Caen
  - CHU de Caen, Caen
  - Hôpitaux Civils de Colmar, Colmar
  - CHRU de Lille, Lille
  - Hôpital la Timone, Marseille
  - CHU Hôpital Gui de Chaulliac, Montpellier
  - CHU Nord - Hôpital Guillaume et René Laënnec, Nantes - Saint Herblain
  - Hôpital Cimiez C.M.R.R., Nice
  - Service d'Imagerie Medicale, Nice
  - Groupe Hospitalier Broca-La Rochefoucauld, Paris
  - Hôpital Pitié-Salpétrière, Paris
  - Hospital Jean Bernard CIC, Poitiers
  - C.H.U de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU - Hopital Charles Nicolle, Rouen
  - Hôpital Purpan, Toulouse
  - CHU Toulouse - Site Casselardit, Toulouse
- Germany (6):
  - Charite-Universitätsmedizin Berlin, Berlin, State of Berlin
  - St. Josef-Klinikum, Bochum
  - Universitaetsklinikum Dresden, Dresden
  - Klinikum der Albert-Ludwigs-Universitaet Freiburg, Freiburg im Breisgau
  - Ortenau Klinikum Offenburg, Offenburg
  - Universitaetsklinikum Ulm, Ulm
- Italy (11):
  - A.O. Umberto I, Ancona
  - Sezione di Neurologia - Dipartimento di Neuroscienze, Ancona
  - Clinica Neurologica - II Neurologia, Brescia
  - Dipartimento di Neuroscienze,, Catania
  - Unita' Operativa Complessa di Neurologia, Catania
  - CeSI (Centro di Scienze dell'invecchiamento) -, Chieti
  - Fondazione IRCCS- Istituto Neurologico Carlo Besta, Milan
  - Ospedale S. Gerardo, Monza
  - Clinica Neurologica, Roma
  - Unita' Operativa C - Riabilitazione Neurologica, Roma
  - Universita degli Studi di Siena, Siena
- Japan (35):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Hospital Organization Tokyo National Hospital, Kiyose, Tokyo
  - Yachiyo Hospital, Aichi
  - Kashiwado Hospital, Chiba
  - National Hospital Organization Chiba-East Hospital, Chiba
  - Nippon Medical School Chiba Hokusoh Hospital, Chiba
  - National Hospital Organization Kokura Medical Center, Fukuoka
  - Maebashi Red Cross Hospital, Gunma
  - Gunma University Hospital, Gunma
  - Shinozuka Hospital, Gunma
  - National Hospital Organization Hiroshima-nishi Medical Ctr., Hiroshima
  - Kobe University Hospital, Hyōgo
  - Nishi-Kobe Medical Center, Hyōgo
  - Kobe City Hospital Org Kobe City Medical Cente West Hp, Hyōgo
  - Kagawa University Hospital, Kagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kanagawa
  - Yokohama City University Medical Center, Kanagawa
  - Shonan Atsugi Hospital, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Minami-Kyoto Hospital, Kyoto
  - National Hospital Organization Maizuru Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Nagano
  - National Hospital Organization Niigata National Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - Okayama University Hospital, Okayama
  - National Hospital Organization Minami-Okayama Medical Center, Okayama
  - Osaka City University Hospital, Osaka
  - Osaka University Hospital, Osaka
  - Kansai Medical University Takii Hospital, Osaka
  - National HP.Org.Shizuoka Inst.Epilepsy,Neurological Disorder, Shizuoka
  - Juntendo University Hospital, Tokyo
  - Juntendo Tokyo Koto Geriatric Medical Center, Tokyo
  - Tokyo Metropolitan Health and Med. Treatment Co. Ebara Hosp, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Mexico (2):
  - OCA Hospital, Monterrey, Nuevo León
  - Instituto Biomedico de Investigacion A.C, Aguascalientes
- Netherlands (9):
  - Amphia Ziekenhuis, Breda, North Brabant
  - Tergooi Ziekenhuizen, Hilversum, North Holland
  - Kennemer Gasthuis, Haarlem, The Netherlands
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Medisch Centrum Alkmaar, Alkmaar
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus MC, Rotterdam
- New Zealand (2):
  - The Memory Clinic, Auckland, NZ
  - Signet Research, Christchurch
- Poland (5):
  - Szpital Uniwersytecki, Oddzial Kliniczny Klinik Chorob Wewnetrznych i, Krakow, Poland
  - NZOZ "NEURO-KARD" "ILKOWSKI I PARTNERZY" Spolka Partnerska Lekarzy, Poznan, Poland
  - NZOZ Dom Suer Ryder, Pallmed Sp. z o.o., Bydgoszcz
  - Oddzial Neurologiczny i Udarowy Szpital Wolski im. dr Anny Gostynskiej,, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Katedra i Klinika, Warsaw
- Portugal (3):
  - Hospital Fernando da Fonseca, Amadora, Amadora
  - Hospitais Da Universidade De Coimbra, Coimbra, Coimbra District
  - Hospital Santa Maria, Lisbon, Lisbon District
- Serbia (5):
  - Klinicki centar Srbije, Belgrade
  - Diagnostic Imaging Center, Kamenitz
  - Institute for Cardiovascular Diseases of Vojvodina, Kamenitz
  - Clinical Centre Kragujevac, Clinic of Psichiatry, Kragujevac
  - Klinicki Centar Vojvodina, Novi Sad
- Slovakia (4):
  - Psychiatricka ambulancia, Bratislava
  - Univerzitna nemocnica Bratislava, Bratislava
  - Psychiatricka nemocnica Michalovce, n.o., Michalovce
  - Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
- South Africa (6):
  - Boithuso Caregivers, Johannesburg, Gauteng
  - The Osteoporosis and Memory Centre, Johannesburg, Gauteng
  - Denmar Clinic, Pretoria, Gauteng
  - St Augustine's Medical Centre 2, Durban, KwaZulu-Natal
  - Flexivest Fourteen Research Center, Bellville, Western Cape
  - Panorama Psychiatry and Memory Clinic, Panorama, Western Cape
- Spain (18):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - CLONUS, Palma de Mallorca, Balearic Islands
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian, Basque Country
  - Hospital Divino Valles, Burgos, Burgos
  - Hospital Virgen del Puerto, Plasencia, Caceres
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de Cruces, Barakaldo, Vizcalla
  - Fundacio ACE Institut Catala de Neurociences Aplicades, Barcelona
  - Centro Internacional de Medicina Avanzda (CIMA), Barcelona
  - Hospital de la Princesa, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
- Sweden (4):
  - Malmo University Hospital, Malmo
  - Uppsala Imanet AB, Uppsala
  - Akademiska Sjukhuset, Uppsala
  - ORKI, enheten for radiologi, Uppsala
- Switzerland (4):
  - Memory Clinic Neuro-Psychologie Zentrum, Basel, Canton of Basel-City
  - Hopitaux Universitaires de Geneve, Les Acacias, Canton of Geneva
  - CHUV Lausanne, Lausanne, Canton of Vaud
  - Hopitaux Universitaires de Geneve, Thonex-Geneva
- United Kingdom (13):
  - Glasgow Memory Clinic, Glasgow, Glasgow
  - MAC UK Neuroscience Ltd, Blackpool, Lancashire
  - Kings College Hospital, London, London
  - MAC UK Neuroscience, Research Assessment Centre, Trafford Park, Manchester
  - Pollard Park Health Centre, Bradford
  - Clinical Investigation and Research Unit (CIRU), Brighton
  - Dept. of Neurosciences Charing Cross Hospital, London
  - Newcastle General Hospital, Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Llandough Hospital, Penarth
  - Royal Hallamshire Hospital, Sheffield
  - Grenoside Grange Hospital, Sheffield
  - Victoria Hospital, Swindon

REFERENCES:
- [Derived] Vandenberghe R, Rinne JO, Boada M, Katayama S, Scheltens P, Vellas B, Tuchman M, Gass A, Fiebach JB, Hill D, Lobello K, Li D, McRae T, Lucas P, Evans I, Booth K, Luscan G, Wyman BT, Hua L, Yang L, Brashear HR, Black RS; Bapineuzumab 3000 and 3001 Clinical Study Investigators. Bapineuzumab for mild to moderate Alzheimer's disease in two global, randomized, phase 3 trials. Alzheimers Res Ther. 2016 May 12;8(1):18. doi: 10.1186/s13195-016-0189-7. PMID 27176461
- [Derived] Lacey L, Bobula J, Rudell K, Alvir J, Leibman C. Quality of Life and Utility Measurement in a Large Clinical Trial Sample of Patients with Mild to Moderate Alzheimer's Disease: Determinants and Level of Changes Observed. Value Health. 2015 Jul;18(5):638-45. doi: 10.1016/j.jval.2015.03.1787. Epub 2015 Apr 10. PMID 26297092
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133K1-3001&StudyName=Study%20Evaluating%20the%20Safety%20and%20Efficacy%20of%20Bapineuzumab%20in%20Alzheimer%20Disease%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 218 centers across the world. The study was terminated early by the sponsor on 06 August 2012. Enrollment had already been completed at the time of this decision. Participants who were still participating at that time were asked to complete an early withdrawal visit.
Groups:
- Placebo: Participants received placebo by intravenous (IV) infusion every 13 weeks up to 6 doses (65 weeks). Participants were followed up until 78 weeks.
- Bapineuzumab: Participants received bapineuzumab 0.5 mg/kg by IV infusion every 13 weeks up to 6 doses (65 weeks). Participants were followed up until 78 weeks
Period: Overall Study
Arm/Group | Placebo | Bapineuzumab
Started | 441 | 658
Treated | 439 | 654
Completed | 285 | 398
Not Completed | 156 | 260
Not completed — Adverse Event | 34 | 60
Not completed — Death | 4 | 4
Not completed — Lack of Efficacy | 0 | 6
Not completed — Lost to Follow-up | 0 | 13
Not completed — Physician Decision | 5 | 8
Not completed — Protocol Violation | 4 | 8
Not completed — Withdrawal by Subject | 24 | 42
Not completed — Discontinuation of study by sponsor | 65 | 88
Not completed — Failed to return | 2 | 1
Not completed — Loss of caregiver | 5 | 3
Not completed — Other | 11 | 20
Not completed — Participant participation unknown | 1 | 4
Not completed — Vasogenic edema recurrence | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one infusion or portion of an infusion of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bapineuzumab | Total
Number analyzed (Participants) | 439 | 654 | 1093
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (7.75) | 71.0 (7.67) | 70.7 (7.71)
Age, Customized [Number; unit: Number of participants]
  <65 years | 97 | 132 | 229
  >=65 years | 342 | 522 | 864
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262 | 421 | 683
  Male | 177 | 233 | 410

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive (ADAS-Cog)/11 Subscale Total Score at Week 78
Description: The ADAS-Cog is a multi-item, objective measure of cognitive function. The scale evaluates memory, language, and praxis with items such as orientation, word recall, word recognition, object identification, comprehension, and the completion of simple tasks. Analysis of the ADAS-Cog for this study was based upon an 11 item score from the following items 1) word recall task, 2) naming objects and fingers, 3) following commands, 4) constructional praxis, 5) ideational praxis, 6) orientation, 7) word recognition, 8) remembering test instructions, 9) spoken language ability, 10) word finding difficulty in spontaneous speech, and 11) comprehension.
  This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced.
  The ADAS-Cog/11 ranged from 0 to 70 points, with higher scores indicating a greater degree of impairment. A negative change from baseline indicates a decrease in cognitive impairment.
Time Frame: Baseline and 78 weeks
Population: The modified intent-to-treat (mITT) included all randomized participants who received at least one infusion or portion of an infusion of study drug and who had a baseline and at least one post-baseline assessment of the ADAS-Cog/11 total score and Disability Assessment for Dementia (DAD) total score.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Groups:
- Placebo: Participants received placebo by IV infusion every 13 weeks up to 6 doses (65 weeks). Participants were followed up until 78 weeks
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 300 | 414
Unit on a scale | 7.31 (0.47) | 7.32 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in ADAS-Cog/11 total score was analyzed using a restricted maximum likelihood-based mixed model for repeated measures. The number of participants in each group gave 90% power to detect a 2.21 point advantage for the bapineuzumab group over placebo on the ADAS-Cog/11 total score, at the primary time point (Week 78). This calculation was based on a two-sided test with an alpha of 0.05; Test type: Superiority or Other; p = 0.979, Mixed Models Analysis — Primary variable ADAS-Cog/11 total score had to reach statistical significance, p-values had to reach p <=0.05, in order to be declared effective; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-1.18 to 1.22]

2. Primary Outcome: Change From Baseline in Disability Assessment for Dementia (DAD) Total Score at Week 78
Description: The DAD measures instrumental and basic activities of daily living in participants with Alzheimer's Disease (AD). The DAD is administered to the participants'caregiver in the form of an interview. This scale had to be administered by a trained and certified psychometric rater who did not have access to any information regarding adverse events experienced by the participant.
  This scale assesses a participants' ability to initiate, plan, and perform activities related to hygiene, dressing, continence, eating, meal preparation, telephoning, going on an outing, finance and correspondence, medications, leisure, and housework. Each item can be scored as 1 = yes, 0 = no, non applicable = NA. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores indicate better function; a positive change from baseline indicates an improvement.
Time Frame: Baseline and 78 weeks
Population: The mITT included all randomized participants who received at least one infusion or portion of an infusion of study drug and who had a baseline and at least one post-baseline assessment of the ADAS-Cog/11 total score and DAD total score.
Measure: Least Squares Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 301 | 411
Unit on a scale | -14.94 (1.00) | -14.89 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in DAD total score was analyzed using a restricted maximum likelihood-based mixed model for repeated measures. The number of participants in each group gave 90% power to detect a 5.39 unit advantage for the bapineuzumab group over placebo on the DAD total score, at the primary time point (Week 78). This calculation was based on a two-sided test with an alpha of 0.05; Test type: Superiority or Other; p = 0.973, Mixed Models Analysis — Primary variable DAD total score had to reach statistical significance, p-values had to reach p <=0.05, in order to be declared effective; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-2.51 to 2.60]

3. Secondary Outcome: Change From Baseline in Brain Amyloid Burden at Week 71
Description: Brain amyloid burden as imaged by 11C-Pittsburgh compound B (PIB) positron emission tomography (PET). The latter is a semi-quantitative measure of the extent of fibrillar amyloid in the brain. PIB PET measurements were made in cortical regions found to have the highest burden of fibrillar amyloid at autopsy in participants diagnosed as having Alzheimer's pathology, and also regions reported to have the highest average retention of PIB signal in previous PET studies enrolling participants with probable AD. This parameter reflects overall brain amyloid deposition as indexed by imaging. The change from baseline was measured as average standard uptake value ratio (SUVr) in prespecified regions of interest (ROI) assessed by PIB PET imaging in a subset of participants.
Time Frame: Baseline and 71 weeks
Population: PIB PET population included all randomized participants who enrolled in the PET substudies and who met the following criteria: a) received at least one infusion or portion of an infusion of study drug, b) had a baseline and at least one postbaseline PIB PET assessment, and c) had an SUVr for the global cortical average (GCA) ROI ≥1.35 at baseline.
Measure: Least Squares Mean (Standard Error); unit: standard uptake value ratio
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 12 | 15
standard uptake value ratio | 0.03 (0.04) | -0.04 (0.03)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in PIB PET SUVr was analyzed using a restricted maximum likelihood-based mixed model for repeated measures. The number of participants gave 90% power to detect a 0.152 unit advantage for the bapineuzumab group over placebo for PiB PET binding at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05; Test type: Superiority or Other; p = 0.159, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.17 to 0.03]

4. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Phospho-tau Levels at Week 71
Description: Biomarkers CSF phospho-tau is an indicator of neuronal injury and neurodegeneration. An elevation in levels of tau, as well as specific p-tau species, is thought to be a marker for progressive cellular degeneration in AD. Accordingly, a reduction from baseline in levels of CSF tau in participants who received bapineuzumab compared with participants who received placebo may be indicative of a reduction in neuronal loss in participants treated with bapineuzumab.
Time Frame: Baseline and 71 Weeks
Population: CSF population included all randomized participants who enrolled in the CSF substudies, received at least one infusion or portion of an infusion of study drug, and had a baseline and at least one postbaseline CSF measurement (CSF phospho-tau).
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 62 | 76
pg/mL | 0.83 (2.04) | -0.55 (1.84)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in CSF phospho-tau was analyzed using an analysis of covariance (ANCOVA) model. The analysis was based on the treatment difference estimated at Week 71 based on appropriate contrasts or LS means. The number of participants gave 90% power to detect a 13-ng/L advantage in phospho-tau for the bapineuzumab group over placebo at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05; Test type: Superiority or Other; p = 0.620, ANCOVA; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-6.89 to 4.13]

5. Secondary Outcome: Change From Baseline in Brain Volume, as Assessed by Magnetic Resonance Imaging Brain Boundary Shift Integral (MRI BBSI), at Week 71
Description: Cerebral atrophy correlates closely with the gradual cognitive decline in AD and can be visualized by MRI. The BBSI technique involves positional matching of serial 3-dimensional MRI brain images, such that brain MRI-image volumes were first registered and then subtracted from each other. Atrophy rates would generally be expected to be lower if the underlying disease was attenuated by effective treatment.
Time Frame: Baseline and 71 Weeks
Population: vMRI population included all randomized participants who enrolled in the vMRI substudies, received at least one infusion or portion of an infusion of study drug, and had a baseline and at least one postbaseline vMRI that passed quality control and was satisfactory for volumetric analysis.
Measure: Least Squares Mean (Standard Error); unit: Milliliter (mL)/year
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 131 | 197
Milliliter (mL)/year | 17.64 (0.69) | 17.51 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in MRI BBSI was analyzed using a restricted maximum likelihood-based mixed model for repeated measures. The number of participants gave 90% power to detect a 4.15-cm3 advantage for the bapineuzumab group over placebo on reduction in brain volume as measured by the BBSI at Week 71. The calculations were based on 2-sided tests with alpha set at 0.05; Test type: Superiority or Other; p = 0.884, Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-1.89 to 1.63]

6. Secondary Outcome: Divergence of Effect on the ADAS-Cog/11 Total Scores From Week 39 to Week 78
Description: Treatment differences are estimated using least-squares (LS) means with factor levels weighted according to overall analysis population proportions. ADAS-Cog/11 total score range is 0 (least impairment) to 70 (most impairment); a negative treatment difference (bapineuzumab minus placebo) favors bapineuzumab. Within the MMRMs for ADAS-Cog/11 described for the primary analyses, linear contrasts were formed to test increasing trend of the differences between bapineuzumab and placebo from Week 39 (the 9-month visit) through Week 78 (the 18 -month visit) for each variable, which is equivalent to testing a positive slope of the differences between each bapineuzumab dose group and placebo from Week 39 through Week 78. Results are from a restricted maximum likelihood (REML)-based mixed model for MMRM.
Time Frame: Week 39 to Week 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units/Year
Groups:
- Bapineuzumab 0.5 mg/kg: Participants received bapineuzumab 0.5 mg/kg by IV infusion every 13 weeks up to 6 doses (65 weeks). Participants were followed up until 78 weeks
Arm/Group | Placebo | Bapineuzumab 0.5 mg/kg
Number analyzed (Participants) | 431 | 650
Units/Year
  Week 39 | 2.95 (0.30) | 2.68 (0.25)
  Week 52 | 4.40 (0.34) | 4.08 (0.29)
  Week 65 | 5.76 (0.39) | 5.16 (0.32)
  Week 78 | 7.31 (0.47) | 7.32 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab 0.5 mg/kg; Treatment Difference: Bapineuzumab - Placebo; Test type: Superiority or Other; p = 0.700, Mixed Models Analysis; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [-0.97 to 1.45]

7. Secondary Outcome: Divergence of Effect on the DAD Total Scores From Week 39 to Week 78
Description: Treatment differences are estimated using least-squares (LS) means with factor levels weighted according to overall analysis population proportions. DAD total score range is 0 to 100; a positive treatment difference (bapineuzumab minus placebo) favors bapineuzumab. Within the MMRMs for ADAS-Cog/11 described for the primary analyses, linear contrasts were formed to test increasing trend of the differences between bapineuzumab and placebo from Week 39 (the 9-month visit) through Week 78 (the 18 -month visit) for each variable, which is equivalent to testing a positive slope of the differences between each bapineuzumab dose group and placebo from Week 39 through Week 78. Results are from a restricted maximum likelihood (REML)-based mixed model for MMRM.
Time Frame: Week 39 to Week 78
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units/Year
Arm/Group | Placebo | Bapineuzumab 0.5 mg/kg
Number analyzed (Participants) | 431 | 650
Units/Year
  Week 39 | -6.60 (0.65) | -6.93 (0.54)
  Week 52 | -9.34 (0.73) | -9.34 (0.61)
  Week 65 | -12.14 (0.91) | -13.04 (0.76)
  Week 78 | -14.94 (1.00) | -14.89 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab 0.5 mg/kg; Treatment Difference: Bapineuzumab - Placebo; Test type: Superiority or Other; p = 0.949, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-2.61 to 2.78]

8. Secondary Outcome: Time to First Median Placebo Deterioration on ADAS-Cog/11 Total Score (European Union [EU] Analysis Plan)
Description: The time to first median placebo deterioration, defined as the first time a participant experienced an increase (worsening) from baseline in ADAS-Cog/11 total score greater than or equal to the median worsening observed at Week 78 in the placebo group. The Kaplan Meier estimate of median time to first median placebo deterioration was presented.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Days | 463.0 [455.0 to 546.0] | 457.0 [455.0 to 541.0]
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.684, Log Rank

9. Secondary Outcome: Time to First Clinically Meaningful Deterioration on ADAS-Cog/11 Total Score (United States [US] Analysis Plan)
Description: The time to first clinically meaningful deterioration was defined as the first time a participant experienced an increase (worsening) from baseline in ADAS-Cog/11 total score of >=7.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Days | NA [546.0 to NA] — Values were not calculable due to the large number of censored event times | 546.0 [546.0 to NA] — Values were not calculable due to the large number of censored event times
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.383, Log Rank

10. Secondary Outcome: Time to First Median Placebo Deterioration on DAD Total Score (EU Analysis Plan)
Description: The time to first median placebo deterioration was defined as the first time a participant experienced a decrease (worsening) in DAD total score greater than or equal to the median worsening at Week 78 in the placebo group.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Days | 464.0 [455.0 to 546.0] | 456.0 [449.0 to 539.0]
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.191, Log Rank

11. Secondary Outcome: Time to First Clinically Meaningful Deterioration on DAD Total Score (US Analysis)
Description: The time to first clinically meaningful deterioration was defined as the first time a participant experienced a decrease (worsening) from baseline in DAD total score of >=12.
Time Frame: Baseline and 78 Weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Days | 546.0 [542.0 to 546.0] | 546.0 [540.0 to 546.0]
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.478, Log Rank

12. Secondary Outcome: Change From Baseline in Dependence Scale Total Score at Week 78
Description: The Dependence Scale (DS) is a 13-item, caregiver-rated instrument for determining the amount of support required by a participant with AD. The DS total score ranges from 0 to 15, with higher scores indicating more need for assistance. The DS was administered as an interview to the caregiver at scheduled study visits.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 316 | 437
Unit on a scale | 1.33 (0.12) | 1.22 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in DS total score was analyzed using a restricted maximum likelihood-based mixed model for repeated measures; Test type: Superiority or Other; p = 0.462, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.41 to 0.13]

13. Secondary Outcome: Percentage of Participants With Worsening From Baseline in ADAS-Cog/11 Total Score at Week 78 (EU Analysis Plan)
Description: Percentage of participants with worsening from baseline to Week 78 in ADAS-Cog/11 total score of ≤0, ≤3, and ≤7 points were reported. In order to calculate time to first median placebo deterioration in ADAS-Cog/11, the median change from baseline to Week 78 among the placebo participants of the mITT analysis population were determined. The median changes were used as the cutpoints for determining "deterioration" for Alzheimer's disease participants in the study. If the median change from baseline to Week 78 in the ADAS-Cog/11 total score among the placebo participants of the mITT Analysis Population is 7 points, then the first median placebo deterioration is the first time where there is a worsening on the ADAS-Cog/11 total score of 7 points or more and the worsening is confirmed by the ADAS-Cog/11 assessment at the next non-missing visit.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Percentage of participants
  Worsening of 0 points | 18.3 [14.8 to 22.3] | 15.5 [12.8 to 18.6]
  Worsening of 3 points | 30.4 [26.1 to 35.0] | 25.5 [22.2 to 29.1]
  Worsening of 7 points | 42.5 [37.7 to 47.3] | 38.0 [34.3 to 41.9]

14. Secondary Outcome: Percentage of Responders for ADAS-Cog/11 Total Score at Week 78 (US Analysis Plan)
Description: Percentage of participants whose increase (worsening) from baseline to Week 78 in ADAS-Cog/11 total score was <7.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Percentage of participant | 42.2 | 37.1
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel

15. Secondary Outcome: Percentage of Participants With Worsening From Baseline in DAD Total Score at Week 78 (EU Analysis Plan)
Description: Percentage of participants whose decrease (worsening) from baseline to Week 78 in DAD total score of ≤ 0, ≤ 6, and ≤ 12 points. In order to calculate time to first median placebo deterioration in DAD, the median change from baseline to Week 78 among the placebo participants of the mITT analysis population were determined. The median changes were used as the cutpoints for determining "deterioration" for Alzheimer's disease participants in the study. If the median change from baseline to Week 78 in the DAD total score among the placebo participants of the mITT Analysis Population is 7 points, then the first median placebo deterioration is the first time where there is a worsening on the DAD total score of 7 points or more and the worsening is confirmed by the DAD assessment at the next non-missing visit.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Percentage of participants
  Worsening of 0 points | 17.2 [13.7 to 21.1] | 18.6 [15.7 to 21.8]
  Worsening of 6 points | 29.9 [25.6 to 34.5] | 27.4 [24.0 to 31.0]
  Worsening of 12 points | 39.7 [35.0 to 44.5] | 34.9 [31.3 to 38.7]

16. Secondary Outcome: Percentage of Responders for DAD Total Score at Week 78 (US Analysis Plan)
Description: Percentage of participants whose decrease (worsening) from baseline to Week 78 in DAD total score was <12.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participant
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 431 | 650
Percentage of participant | 39.7 | 34.9
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Test type: Superiority or Other; p = 0.120, Cochran-Mantel-Haenszel

17. Secondary Outcome: Change From Baseline in Clinical Dementia Rating Sum of Boxes (CDR-SOB) Total Score at Week 78
Description: The CDR-SOB is a global clinical staging instrument that sums 6 clinical ratings: 1) memory, 2) orientation, 3) judgment and problem solving, 4) involvement in community affairs, 5) home and hobbies, and 6) personal care based on the Clinical Dementia Rating Scale (CDR) interview. The CDR includes discussions with the participant and caregiver using a structured format. This scale had to be administered by a trained and certified global rater who did not have access to any information regarding adverse events experienced by the participant. CDR-SOB total score range is 0 (least impairment) to 18 (most impairment); a negative change from baseline indicates an improvement.
Time Frame: Baseline and 78 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Bapineuzumab
Number analyzed (Participants) | 310 | 427
Units on a scale | 2.59 (0.16) | 2.44 (0.13)
Statistical Analysis 1: Comparison: Placebo vs Bapineuzumab; Change in CDR-SOB total score was analyzed using a restricted maximum likelihood-based mixed model for repeated measures; Test type: Superiority or Other; p = 0.448, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.55 to 0.24]

ADVERSE EVENTS:
Time Frame: 4 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Bapineuzumab
Serious Adverse Events (participants affected / at risk) | 77/439 | 137/654
Other Adverse Events (participants affected / at risk) | 198/439 | 298/654
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=439) | Bapineuzumab (N=654)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2)
Device occlusion (General disorders) | 0 (0) | 1 (1)
Fibrosis (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Bacterial Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 6 (6)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (4) | 1 (1)
Toxic shock syndrome (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vaginitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (5)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (5) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (7) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (5) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Streptococcus test positive (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (5)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral haemosiderin deposition (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 4 (4)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (3)
Lacunar infarction (Nervous system disorders) | 1 (4) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Mental impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 4 (4)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 4 (5) | 40 (61)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 1 (3) | 2 (2)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 3 (3)
Delirium (Psychiatric disorders) | 1 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2) | 3 (3)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Social problem (Social circumstances) | 0 (0) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 5 (5)
Ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=439) | Bapineuzumab (N=654)
Diarrhoea (Gastrointestinal disorders) | 23 (30) | 34 (38)
Nasopharyngitis (Infections and infestations) | 34 (40) | 45 (66)
Urinary tract infection (Infections and infestations) | 24 (37) | 30 (34)
Fall (Injury, poisoning and procedural complications) | 27 (36) | 39 (47)
Cerebral microhaemorrhage (Nervous system disorders) | 16 (38) | 76 (218)
Dizziness (Nervous system disorders) | 23 (32) | 20 (26)
Headache (Nervous system disorders) | 44 (98) | 45 (66)
Vasogenic cerebral oedema (Nervous system disorders) | 5 (5) | 74 (123)
Anxiety (Psychiatric disorders) | 26 (29) | 30 (61)
Depression (Psychiatric disorders) | 27 (73) | 35 (95)
Hypertension (Vascular disorders) | 22 (50) | 18 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.